CLINICAL TRIAL: NCT00227877
Title: Screening and Brief Advice to Reduce Teen Substance Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Cambridge Health Alliance (Other); Concord Hospital (Other); Fallon Clinic (Industry); Tufts Medical Center (Other); University of Vermont (Other)
Responsible Party: Principal Investigator, John R Knight, MD, Associate Professor of Pediatrics, Harvard Medical School, Boston Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIDA-R01DA0118848; NCT00592878 (obsolete NCT alias); NCT00592956 (obsolete NCT alias)
Record Dates: First submitted 2005-09-27; First posted 2005-09-28 (Estimated); Results first posted 2018-09-21 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Substance Related Disorders
Keywords: alcohol abuse; substance abuse; substance related disorders
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism

STUDY DESIGN:
Intervention Model Description: In this before-/after- quasi-experimental trial, all sites first completed a treatment-as-usual phase with assessments only, followed by all sites undergoing training and completing a subsequent intervention phase.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control - New England, USA (No Intervention): Control participants will receive "care as usual" from their provider
- cSBA - New England, USA (Experimental): Participants who are in the experimental arm will complete the CRAFFT screen on the computer and receive information on the computer regarding the health effects of substance use. Their provider will be given the results of their CRAFFT screen and a list of suggested "talking points" which they will use to guide a discussion with the patient about drug and alcohol use. Participants and their families will also receive educational brochures about substance use.
  Interventions: Behavioral: cSBA - New England, USA
- Control - Prague, CZR (No Intervention): Control participants will receive "care as usual" from their provider
- cSBA - Prague, CZR (Experimental): Participants who are in the experimental arm will complete the CRAFFT screen on the computer and receive information on the computer regarding the health effects of substance use. Their provider will be given the results of their CRAFFT screen and a list of suggested "talking points" which they will use to guide a discussion with the patient about drug and alcohol use. Participants and their families will also receive educational brochures about substance use.
  Interventions: Behavioral: cSBA - Prague, CZR

INTERVENTIONS:
Behavioral: cSBA - New England, USA — Participants who are in the experimental arm will complete the CRAFFT screen on the computer and receive information on the computer regarding the health effects of substance use. Their provider will be given the results of their CRAFFT screen and a list of suggested "talking point" which they will use to guide a discussion with the patient about drug and alcohol use. Participants and their families will also receive educational brochures about substance use.
  Other Names: SBIRT
  Arms: cSBA - New England, USA
Behavioral: cSBA - Prague, CZR — Participants who are in the experimental arm will complete the CRAFFT screen on the computer and receive information on the computer regarding the health effects of substance use. Their provider will be given the results of their CRAFFT screen and a list of suggested "talking point" which they will use to guide a discussion with the patient about drug and alcohol use. Participants and their families will also receive educational brochures about substance use.
  Other Names: SBIRT
  Arms: cSBA - Prague, CZR

SUMMARY:
The purpose of this study is to test the effectiveness of a brief intervention for alcohol and drug use in adolescents that a primary care doctor can give in his/her office. The study will be conducted in nine primary care offices in three New England states, and in ten pediatric offices in Prague, Czech Republic (CZR).

We hypothesize that:

1. Among 12-18 year old well care patients who screen positive for drug/alcohol use, the experimental intervention administered by trained primary care providers will be more effective than standard care in decreasing drug and alcohol use;
2. Among 12-18 year old well care patients who screen negative for drug/alcohol use, the experimental intervention administered by trained primary care providers will be more effective than standard care in decreasing initiation of drug and alcohol use as measured by self-reports of substance use;
3. Among 12-18 year old well care patients who are at risk for riding with an impaired driver or driving while impaired, the experimental intervention administered by trained primary care providers will be more effective than standard care in decreasing Riding/Driving risk behavior as measured by a standardized scale.

DETAILED DESCRIPTION:
We are trying to find out the best way for doctors to talk with their adolescent patients about alcohol and drug use. Adolescents 12-18 who are coming to their doctor's office for a routine well-care or follow-up visit will be invited to participate in the study. Participants do not have to have ever used alcohol or drugs. All participants will answer a computerized questionnaire about alcohol and drug use three times. The first one will be at the time of a doctor's visit. The second time will be three months later and the third time a year later. Adolescents who agree to be in the study during the first year will be in the 'control' group. Their doctor will talk to them about drugs and alcohol the same as he/she usually does for all his/her patients. Those who agree to be in the study during the second year will be in the 'intervention' group. Everyone in the 'intervention' group will receive some advice on the computer about their alcohol and drug use. Their doctor will also give them some specific advice about drug and alcohol use. The researchers have chosen what that advice will be, and all doctors involved in the study will give advice according to the study protocol. Participants and their parents will also be given educational information about alcohol and drugs. We will test the effectiveness of the intervention by comparing drug and alcohol use between those who are in the 'control' group, and those who are in the 'intervention' group.

We we will also validate the Czech version of the CRAFFT screen before conducting the effectiveness trial outlined above in the Czech Republic.

ELIGIBILITY:
Inclusion Criteria:

12-18 year old patients coming for well care or follow-up visits to one of the study sites, All levels of substance use, Able to read and understand English

Exclusion Criteria:

Will not be available for 12 month follow-up period, Medically unstable at the time of the visit

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2695 (Actual)
Dates: Start 2005-12 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R Knight, M.D., Principal Investigator — Boston Children's Hospital
Locations (6):
- United States (5):
  - Tufts-New England Medical Center, Boston, Massachusetts
  - Cambridge Pediatrics, Cambridge, Massachusetts
  - Fallon Clinic, Worcester, Massachusetts
  - Capital Region Family Health Center, Concord, New Hampshire
  - Milton Family Practice, Milton, Vermont
- Center for the Evaluation, Prevention, and Research of Substance Abuse, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knight JR, Shrier LA, Bravender TD, Farrell M, Vander Bilt J, Shaffer HJ. A new brief screen for adolescent substance abuse. Arch Pediatr Adolesc Med. 1999 Jun;153(6):591-6. doi: 10.1001/archpedi.153.6.591. PMID 10357299
- [Background] Knight JR, Sherritt L, Shrier LA, Harris SK, Chang G. Validity of the CRAFFT substance abuse screening test among adolescent clinic patients. Arch Pediatr Adolesc Med. 2002 Jun;156(6):607-14. doi: 10.1001/archpedi.156.6.607. PMID 12038895
- [Background] Van Hook S, Harris SK, Brooks T, Carey P, Kossack R, Kulig J, Knight JR; New England Partnership for Substance Abuse Research. The "Six T's": barriers to screening teens for substance abuse in primary care. J Adolesc Health. 2007 May;40(5):456-61. doi: 10.1016/j.jadohealth.2006.12.007. Epub 2007 Feb 15. PMID 17448404
- [Background] Knight JR, Harris SK, Sherritt L, Van Hook S, Lawrence N, Brooks T, Carey P, Kossack R, Kulig J. Prevalence of positive substance abuse screen results among adolescent primary care patients. Arch Pediatr Adolesc Med. 2007 Nov;161(11):1035-41. doi: 10.1001/archpedi.161.11.1035. PMID 17984404
- [Background] Knight JR, Harris SK, Sherritt L, Van Hook S, Lawrence N, Brooks T, Carey P, Kossack R, Kulig J. Adolescents' preference for substance abuse screening in primary care practice. Subst Abus. 2007;28(4):107-17. doi: 10.1300/J465v28n04_03. PMID 18077307
- [Result] Knight JR, Csemy L, Sherritt L, Starostova O, Van Hook S, Bacic J, Finlay C, Tauber J, Brooks T, Kossack R, Kulig JW, Shaw J, Harris SK. Screening and Brief Advice to Reduce Adolescents' Risk of Riding With Substance-Using Drivers. J Stud Alcohol Drugs. 2018 Jul;79(4):611-616. doi: 10.15288/jsad.2018.79.611. PMID 30079877
- [Result] Knight JR, Kuzubova K, Csemy L, Sherritt L, Copelas S, Harris SK. Computer-Facilitated Screening and Brief Advice to Reduce Adolescents' Heavy Episodic Drinking: A Study in Two Countries. J Adolesc Health. 2018 Jan;62(1):118-120. doi: 10.1016/j.jadohealth.2017.08.013. Epub 2017 Oct 17. PMID 29054734
- [Result] Hadland SE, Copelas SH, Harris SK. Trajectories of Substance Use Frequency among Adolescents Seen in Primary Care: Implications for Screening. J Pediatr. 2017 May;184:178-185. doi: 10.1016/j.jpeds.2017.01.033. Epub 2017 Feb 10. PMID 28196680
- [Result] Harris SK, Johnson JK, Sherritt L, Copelas S, Rappo MA, Wilson CR. Putting Adolescents at Risk: Riding With Drinking Drivers Who Are Adults in the Home. J Stud Alcohol Drugs. 2017 Jan;78(1):146-151. doi: 10.15288/jsad.2017.78.146. PMID 27936375
- [Result] Louis-Jacques J, Knight JR, Sherritt L, Van Hook S, Harris SK. Do risky friends change the efficacy of a primary care brief intervention for adolescent alcohol use? J Adolesc Health. 2014 Apr;54(4):449-53. doi: 10.1016/j.jadohealth.2013.09.012. Epub 2013 Nov 8. PMID 24216313
- [Result] Harris SK, Csemy L, Sherritt L, Starostova O, Van Hook S, Johnson J, Boulter S, Brooks T, Carey P, Kossack R, Kulig JW, Van Vranken N, Knight JR. Computer-facilitated substance use screening and brief advice for teens in primary care: an international trial. Pediatrics. 2012 Jun;129(6):1072-82. doi: 10.1542/peds.2011-1624. Epub 2012 May 7. PMID 22566420
- [Derived] Byregowda H, Flynn AL, Knight JR, Harris SK. Perceived Risk of Harm Mediates the Effects of Primary Care Alcohol Use Screening and Brief Advice in Adolescents. J Adolesc Health. 2022 Mar;70(3):442-449. doi: 10.1016/j.jadohealth.2021.09.029. Epub 2021 Dec 31. PMID 34974918
- [Derived] Knight JR, Sherritt L, Gibson EB, Levinson JA, Grubb LK, Samuels RC, Silva T, Vernacchio L, Wornham W, Harris SK. Effect of Computer-Based Substance Use Screening and Brief Behavioral Counseling vs Usual Care for Youths in Pediatric Primary Care: A Pilot Randomized Clinical Trial. JAMA Netw Open. 2019 Jun 5;2(6):e196258. doi: 10.1001/jamanetworkopen.2019.6258. PMID 31225897
- See also: This is the web site of the Center for Adolescent Substance Use and Addiction Research (CeASAR) at Children's Hospital Boston. CeASAR is the research center funded to direct this project. — http://www.crafft.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Quasi-experimental, asynchronous study design with each site as its own control. From 2005 to 2008, 12- to 18-year-olds arriving for routine care at 9 medical offices in New England (n= 2096, 58% females) and 10 in Prague, Czech Republic (n = 589, 47% females) were recruited. Medically/emotionally stable, able to read, and available for follow-ups.
Groups:
- Control - New England; Control - Czech Republic: Control participants received "care as usual" from their provider
- cSBA - New England: Computer screen & brief physician advice: Participants in the experimental arm completed a computerized CRAFFT screen and received information on the computer regarding the health effects of substance use. Their provider was given the results of their CRAFFT screen and a list of suggested "talking points" which guided a discussion with the patient about drug and alcohol use.
- cSBA - Czech Republic: Computer screen & brief physician advice: Participants in the experimental arm completed a computerized CRAFFT screen and received information on the computer regarding the health effects of substance use. Their provider was given the results of their CRAFFT screen and a list of suggested "talking points" to guide a discussion with the patient about drug and alcohol use.
Period: Pre-visit Assessment
Arm/Group | Control - New England | cSBA - New England | Control - Czech Republic | cSBA - Czech Republic
Started | 1075 | 1031 | 297 | 292
Completed | 1068 (Final analysis sample) | 1028 (Final analysis sample) | 297 (Final analysis sample) | 292 (Final analysis sample)
Not Completed | 7 | 3 | 0 | 0
Not completed — Technical difficulties | 7 | 3 | 0 | 0
Period: Post-visit Checklist
Arm/Group | Control - New England | cSBA - New England | Control - Czech Republic | cSBA - Czech Republic
Started | 1068 | 1028 | 297 | 292
Completed | 1044 | 1015 | 296 | 292
Not Completed | 24 | 13 | 1 | 0
Not completed — Lost to Follow-up | 24 | 13 | 1 | 0
Period: 3-months Follow-up
Arm/Group | Control - New England | cSBA - New England | Control - Czech Republic | cSBA - Czech Republic
Started (These "Started" numbers reflect those who completed the pre-visit assessment.) | 1068 | 1028 | 297 | 292
Completed | 755 | 761 | 245 | 271
Not Completed | 313 | 267 | 52 | 21
Not completed — Completed late | 135 | 128 | 34 | 8
Not completed — Lost to Follow-up | 178 | 139 | 18 | 13
Period: 12-months Follow-up
Arm/Group | Control - New England | cSBA - New England | Control - Czech Republic | cSBA - Czech Republic
Started (These "Started" numbers reflect those who completed the pre-visit assessment.) | 1068 | 1028 | 297 | 292
Completed | 758 | 765 | 266 | 266
Not Completed | 310 | 263 | 31 | 26
Not completed — Completed late | 78 | 74 | 1 | 0
Not completed — Lost to Follow-up | 232 | 189 | 30 | 26

BASELINE CHARACTERISTICS:
Groups:
- Control - New England; Control - Czech Republic: Control participants will receive "care as usual" from their provider
- Computer Screen & Brief Physician Advice - New England; Computer Screen & Brief Physician Advice - Czech Republic: Participants who are in the experimental arm will complete the CRAFFT screen on the computer and receive information on the computer regarding the health effects of substance use. Their provider will be given the results of their CRAFFT screen and a list of suggested "talking points" which they will use to guide a discussion with the patient about drug and alcohol use. Participants and their families will also receive educational brochures about substance use.
  Computer screen & brief physician advice: Participants who are in the experimental arm will complete the CRAFFT screen on the computer and receive information on the computer regarding the health effects of substance use. Their provider will be given the results of their CRAFFT screen and a list of suggested "talking point" which they will use to guide a discussion with the patient about drug and alcohol use. Participants and their families will also receive educational brochures about substance use.
- Total: Total of all reporting groups
Arm/Group | Control - New England | Computer Screen & Brief Physician Advice - New England | Control - Czech Republic | Computer Screen & Brief Physician Advice - Czech Republic | Total
Number analyzed (Participants) | 1068 | 1028 | 297 | 292 | 2685
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 7 participants removed due to technical difficulties in Control group; 3 participants removed due to technical difficulties in cSBA intervention group
  years
    Age | 15.9 (2.0) | 15.6 (2.0) | 15.0 (1.6) | 15.0 (1.6) | 15.8 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 659 | 561 | 139 | 139 | 1498
  Male | 409 | 467 | 158 | 153 | 1187
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-Hispanic | 689 | 664 | 297 | 292 | 1942
  Hispanic | 106 | 124 | 0 | 0 | 230
  Asian non-Hispanic | 77 | 74 | 0 | 0 | 151
  Black non-Hispanic | 100 | 117 | 0 | 0 | 217
  Other non-Hispanic | 96 | 49 | 0 | 0 | 145
Parents at Home [Count of Participants; unit: Participants] — Population: Number analyzed in three study arm columns for this measure differs from overall number of baseline participants due to missing data on these characteristics for several participants in these arms.
  Participants
    number analyzed (Participants) | 1044 | 1015 | 291 | 292 | 2642
    Two parents | 703 | 721 | 184 | 195 | 1803
    One parent or Other | 341 | 294 | 107 | 97 | 839
Parents Highest Education Level [Count of Participants; unit: Participants] — Population: Number analyzed in the study arm columns for this measure differs from overall number of baseline participants due to missing data on these characteristics for several participants in these arms.
  Participants
    number analyzed (Participants) | 1023 | 1002 | 290 | 290 | 2605
    College/university degree or higher | 451 | 522 | 92 | 100 | 1165
    High school/Secondary school graduate | 427 | 405 | 111 | 106 | 1049
    Did not complete high school/secondary school | 46 | 33 | 44 | 46 | 169
    Don't know | 99 | 42 | 43 | 38 | 222
Visit type [Count of Participants; unit: Participants] — Population: Number analyzed in the study arm columns for this measure differs from overall number of baseline participants due to missing data on these characteristics for several participants in these arms.
  Participants
    Well visit: number analyzed (Participants) | 1050 | 1019 | 297 | 292 | 2658
    Well visit: Yes | 851 | 968 | 297 | 292 | 2408
    Well visit: No | 199 | 51 | 0 | 0 | 250
    First visit: number analyzed (Participants) | 1045 | 1019 | 0 | 0 | 2064
    First visit: Yes | 115 | 105 | 0 | 0 | 220
    First visit: No | 930 | 914 | 0 | 0 | 1844
    Female provider: number analyzed (Participants) | 1054 | 1019 | 296 | 292 | 2661
    Female provider: Yes | 663 | 684 | 263 | 259 | 1869
    Female provider: No | 391 | 335 | 33 | 33 | 792
Parent Substance Use [Count of Participants; unit: Participants] — Population: Number analyzed in the study arm columns for this measure differs from overall number of baseline participants due to missing data on these characteristics for several participants in these arms.
  Participants
    number analyzed (Participants) | 1068 | 1027 | 297 | 292 | 2684
    (all) | 170 | 152 | 32 | 32 | 386
Sibling Substance Abuse [Count of Participants; unit: Participants] | 205 | 187 | 41 | 36 | 469
Peer substance abuse [Count of Participants; unit: Participants] — Population: Number analyzed in the study arm columns for this measure differs from overall number of baseline participants due to missing data on these characteristics for several participants in these arms.
  Participants
    number analyzed (Participants) | 1065 | 1027 | 296 | 292 | 2680
    (all) | 658 | 607 | 204 | 192 | 1661

OUTCOME MEASURES:

1. Primary Outcome: Past-90-day Substance Use at 3 Months Among Baseline Substance Users - New England, USA
Description: Among the 12-18 year old primary care patients who reported past-12-month drug or alcohol use at baseline in New England, USA, this analysis reports the number who subsequently reported past-90-day drug or alcohol use at the 3 months post-baseline assessment.
Time Frame: Past-90-days at 3 months post-baseline
Population: 12-18 year old primary care patients who report past-12-month drug or alcohol use at baseline in New England, USA
Measure: Count of Participants; unit: Participants
Groups:
- Control - New England, USA: Control participants received "care as usual" from their providers
- Computer Screen & Brief Physician Advice - New England, USA: Participants in the experimental arm completed the CRAFFT screen on the computer and received information on the computer regarding the health effects of substance use. Their providers were given the results of their CRAFFT screen and a list of suggested "talking points" which they used to guide a discussion with the patient about drug and alcohol use. Participants and their families also received educational brochures about substance use.
Arm/Group | Control - New England, USA | Computer Screen & Brief Physician Advice - New England, USA
Number analyzed (Participants) | 260 | 222
Participants | 162 | 121
Statistical Analysis 1: Comparison: Control - New England, USA vs Computer Screen & Brief Physician Advice - New England, USA; Test type: Superiority; p < 0.05, Regression, Logistic; Group Conditional Risk Ratio adjusting for the multi-site sample design using GEE logistic regression (SUDAAN 10.0); Adjusted Relative Risk Ratio = 1.39, 95% CI 2-sided [1.08 to 1.80], Standard Error of Mean .18 — Risk Ratio: (Intervention Cessation)/(Control Cessation) controlling for age; gender; parent education; number of parents in home; visit type; perceived parent, sibling, and peer substance use; provider gender; and connectedness to provider

2. Primary Outcome: Past-90-day Substance Use at 3 Months Among Baseline Substance Non-Users, New England, USA
Description: Among the 12-18 year old primary care patients who did NOT report past-12-month drug or alcohol use at baseline in New England, USA, this analysis reports the number who subsequently reported past-90-day drug or alcohol use at the 3 months post-baseline assessment.
Time Frame: Past-90-days at 3 months post-baseline
Population: 12-18 year old primary care patients who did not report past-12-month drug or alcohol use at baseline in New England, USA
Measure: Count of Participants; unit: Participants
Groups:
- Control - New England, USA: Control participants received "care as usual" from their provider
- cSBA - New England, USA: Computer Screen & Brief physician Advice: Participants in the experimental arm completed a computerized CRAFFT screen and received information on the computer regarding the health effects of substance use. Their provider was given the results of their CRAFFT screen and a list of suggested "talking points" which guided a discussion with the patient about drug and alcohol use.
Arm/Group | Control - New England, USA | cSBA - New England, USA
Number analyzed (Participants) | 494 | 539
Participants | 24 | 15
Statistical Analysis 1: Comparison: Control - New England, USA vs cSBA - New England, USA; Test type: Superiority; p = .32, Regression, Logistic; Group Conditional Risk Ratio adjusting for the multi-site sample design using GEE logistic regression (SUDAAN 10.0); Adjusted Relative Risk Ratio = 0.70, 95% CI 2-sided [0.34 to 1.42], Standard Error of Mean 0.25 — Risk Ratio: (Intervention Initiation)/(Control Initiation) controlling for age; gender; parent education; number of parents in home; visit type; perceived parent, sibling, and peer substance use; provider gender; and connectedness to provider

3. Primary Outcome: Past-12-month Substance Use at 12 Months Among Baseline Substance Users, New England, USA
Description: Of those participants who reported past-12-month drug or alcohol use at baseline,the number reporting past-90-day drug or alcohol use at 12 months post-baseline assessment in New England, USA
Time Frame: Past-12-months at 12 months post-baseline
Population: 12-18 year old primary care patients who reported past-12-month drug or alcohol use at baseline in New England, USA
Measure: Count of Participants; unit: Participants
Arm/Group | Control - New England, USA | Computer Screen & Brief Physician Advice - New England, USA
Number analyzed (Participants) | 257 | 209
Participants | 214 | 172
Statistical Analysis 1: Comparison: Control - New England, USA vs Computer Screen & Brief Physician Advice - New England, USA; Test type: Superiority; p = 0.05, Regression, Logistic; Group Conditional Risk Ratio adjusting for the multi-site sample design using GEE logistic regression (SUDAAN 10.0); Adjusted Relative Risk Ratio = 1.80, 95% CI 2-sided [.99 to 3.27], Standard Error of Mean 0.55; Risk Ratio: (Intervention Cessation)/(Control Cessation) controlling for age; gender; parent education; number of parents in home; visit type; perceived parent, sibling, and peer substance use; provider gender; and connectedness to provider

4. Primary Outcome: Past-12-month Substance Use at 12 Months, Baseline Substance Non-Users, New England, USA
Description: Of those participants who reported NO past-12-month drug or alcohol use at baseline,the number reporting past-90-day drug or alcohol use at 12 months post-baseline assessment in New England, USA
Time Frame: Past-12-months at 12 months post-baseline
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Control - New England, USA | cSBA - New England, USA
Number analyzed (Participants) | 500 | 556
Participants | 83 | 73
Statistical Analysis 1: Comparison: Control - New England, USA vs cSBA - New England, USA; Test type: Superiority; p = 0.23, Regression, Logistic; Group Conditional Risk Ratio adjusting for the multi-site sample design using GEE logistic regression (SUDAAN 10.0); Adjusted Relative Risk Ratio = .79, 95% CI 2-sided [.53 to 1.16], Standard Error of Mean .16 — [estimate comment as in outcome 2, analysis 1]

5. Primary Outcome: Past-90-day Substance Use at 3 Months Among Baseline Substance Users - Prague, CZR
Description: Of those participants who reported past-12-month drug or alcohol use at baseline,the number reporting past-90-day drug or alcohol use at 3 months post-baseline assessment in Prague, Czech Republic
Time Frame: Past-90-days at 3 months post-baseline
Population: 12-18 year old primary care patients who reported past-12-month drug or alcohol use at baseline in Prague, CZR
Measure: Count of Participants; unit: Participants
Groups:
- Control - Prague, CZR: Control participants received "care as usual" from their provider
- cSBA - Prague, CZR: Computer Screen & Brief physician Advice: Participants in the experimental arm completed a computerized CRAFFT screen and received information on the computer regarding the health effects of substance use. Their provider was given the results of their CRAFFT screen and a list of suggested "talking points" which guided a discussion with the patient about drug and alcohol use.
Arm/Group | Control - Prague, CZR | cSBA - Prague, CZR
Number analyzed (Participants) | 157 | 161
Participants | 118 | 114
Statistical Analysis 1: Comparison: Control - Prague, CZR vs cSBA - Prague, CZR; Test type: Superiority; p = .07, Regression, Logistic; Group Conditional Risk Ratio adjusting for the multi-site sample design using GEE logistic regression (SUDAAN 10.0); Adjusted Relative Risk Ratio = 1.52, 95% CI 2-sided [.97 to 2.36], Standard Error of Mean 0.34 — Risk Ratio: (Intervention Cessation)/(Control Cessation) controlling for age and gender

6. Primary Outcome: Past-90-day Substance Use at 3 Months Among Baseline Substance Non-Users - Prague, CZR
Description: Of those participants who reported NO past-12-month drug or alcohol use at baseline,the number reporting past-90-day drug or alcohol use at 3 months post-baseline assessment in Prague, Czech Republic
Time Frame: Past-90-days at 3 months post-baseline
Population: 12-18 year old primary care patients who did not report past-12-month drug or alcohol use at baseline in Prague, CZR
Measure: Count of Participants; unit: Participants
Arm/Group | Control - Prague, CZR | cSBA - Prague, CZR
Number analyzed (Participants) | 88 | 110
Participants | 10 | 13
Statistical Analysis 1: Comparison: Control - Prague, CZR vs cSBA - Prague, CZR; Test type: Superiority; p = .93, Regression, Logistic; Adjusted Relative Risk Ratio = .96, 95% CI 2-sided [.42 to 2.21], Standard Error of Mean .41 — Risk Ratio: (Intervention Initiation)/(Control Initiation) controlling for age and gender

7. Primary Outcome: Past-12-Month Substance Use at 12 Months Among Baseline Substance Users - Prague, CZR
Description: Of those participants who reported past-12-month drug or alcohol use at baseline,the number reporting past-12-month drug or alcohol use at 12 months post-baseline assessment in Prague, Czech Republic
Time Frame: Past-12-months at 12 months post-baseline
Population: 12-18 year old primary care patients who reported past-12-month drug or alcohol use at baseline in Prague, CZR
Measure: Count of Participants; unit: Participants
Arm/Group | Control - Prague, CZR | cSBA - Prague, CZR
Number analyzed (Participants) | 163 | 153
Participants | 154 | 148
Statistical Analysis 1: Comparison: Control - Prague, CZR vs cSBA - Prague, CZR; Test type: Superiority; p = .78, Regression, Logistic; Group Conditional Risk Ratio adjusting for the multi-site sample design using GEE logistic regression (SUDAAN 10.0); Adjusted Relative Risk Ratio = .85, 95% CI 2-sided [.27 to 2.70], Standard Error of Mean .50 — Risk Ratio: (Intervention Cessation)/(Control Cessation) controlling for age and gender

8. Primary Outcome: Past-12-Month Substance Use at 12 Months Among Baseline Substance Non-Users - Prague, CZR
Description: as for outcome 7
Time Frame: Past-12-months at 12 months post-baseline
Population: 12-18 year old primary care patients who did not report past-12-month drug or alcohol use at baseline in Prague, CZR
Measure: Count of Participants; unit: Participants
Arm/Group | Control - Prague, CZR | cSBA - Prague, CZR
Number analyzed (Participants) | 103 | 111
Participants | 48 | 38
Statistical Analysis 1: Comparison: Control - Prague, CZR vs cSBA - Prague, CZR; Test type: Superiority; p = .13, Regression, Logistic; Group Conditional Risk Ratio adjusting for the multi-site sample design using GEE logistic regression (SUDAAN 10.0); Adjusted Relative Risk Ratio = .74, 95% CI 2-sided [.51 to 1.09], Standard Error of Mean .15 — Risk Ratio: (Intervention Initiation)/(Control Initiation) controlling for age and gender

9. Secondary Outcome: Any Risky Riding or Driving at 3 Months - New England, USA
Description: Any past-90-day self-reported Riding with a driver who had used alcohol or other drugs or Driving after having used alcohol or other drugs at 3 months post-baseline assessment - New England
Time Frame: Past-90-days at 3 months post-baseline
Population: 12-18 year old primary care patients in New England, USA
Measure: Count of Participants; unit: Participants
Arm/Group | Control - New England, USA | cSBA - New England, USA
Number analyzed (Participants) | 754 | 758
Participants | 150 | 88
Statistical Analysis 1: Comparison: Control - New England, USA vs cSBA - New England, USA; Test type: Superiority; p = .66, Regression, Logistic; Group Conditional Risk Ratio adjusting for the multi-site sample design using GEE logistic regression (SUDAAN 10.0); Adjusted Relative Risk Ratio = .66, 95% CI 2-sided [.48 to .91], Standard Error of Mean .11 — Risk Ratio: (Intervention)/(Control) controlling for age; gender; parent education; number of parents in home; visit type; provider gender; connectedness to provider, and baseline DRWI risk

10. Secondary Outcome: Any Risky Riding or Driving at 12 Months - New England, USA
Description: Any past-90-day self-reported Riding with a driver who had used alcohol or other drugs or Driving after having used alcohol or other drugs at 12 months post-baseline assessment - New England
Time Frame: Past-90-days at 12 months post-baseline
Population: 12-18 year old primary care patients in New England, USA
Measure: Count of Participants; unit: Participants
Arm/Group | Control - New England, USA | cSBA - New England, USA
Number analyzed (Participants) | 756 | 765
Participants | 161 | 125
Statistical Analysis 1: Comparison: Control - New England, USA vs cSBA - New England, USA; Test type: Superiority; p = .35, Regression, Logistic — Group Conditional Risk Ratio adjusting for the multi-site sample design using GEE logistic regression (SUDAAN 10.0); Adjusted Relative Risk Ratio = .87, 95% CI 2-sided [.64 to 1.17], Standard Error of Mean .13 — [estimate comment as in outcome 9, analysis 1]

11. Secondary Outcome: Any Risky Riding or Driving at 3 Months - Prague, CZR
Description: Any past-90-day self-reported Riding with a driver who had used alcohol or other drugs or Driving after having used alcohol or other drugs at 3 months post-baseline assessment - Prague, Czech Republic
Time Frame: Past-90-days at 3 months post-baseline
Population: 12-18 year old primary care patients in Prague, CZR
Measure: Count of Participants; unit: Participants
Arm/Group | Control - Prague, CZR | cSBA - Prague, CZR
Number analyzed (Participants) | 245 | 269
Participants | 245 | 269
Statistical Analysis 1: Comparison: Control - Prague, CZR vs cSBA - Prague, CZR; Test type: Superiority; p < .01, Regression, Logistic; Adjusted Relative Risk Ratio = .63, 95% CI 2-sided [.46 to .87], Standard Error of Mean .10 — Risk Ratio: (Intervention)/(Control) controlling for age; gender; connectedness to provider, and baseline DRWI risk

12. Secondary Outcome: Any Risky Riding or Driving at 12 Months - Prague, CZR
Description: Any past-90-day self-reported Riding with a driver who had used alcohol or other drugs or Driving after having used alcohol or other drugs at 12 months post-baseline assessment - Prague, Czech Republic
Time Frame: Past-90-days at 12 months post-baseline
Population: 12-18 year old primary care patients in Prague, CZR
Measure: Count of Participants; unit: Participants
Arm/Group | Control - Prague, CZR | cSBA - Prague, CZR
Number analyzed (Participants) | 266 | 263
Participants | 78 | 61
Statistical Analysis 1: Comparison: Control - Prague, CZR vs cSBA - Prague, CZR; Test type: Superiority; p < 0.05, Regression, Logistic; Adjusted Relative Risk Ratio = .73, 95% CI 2-sided [.54 to .98], Standard Error of Mean .11 — Risk Ratio: (Intervention)/(Control) controlling for age; gender; connectedness to provider, and baseline DRWI risk

ADVERSE EVENTS:
Time Frame: Through the course of the entire recruitment and follow-up period.
Arm/Group | Control - New England | Computer Screen & Brief Physician Advice - New England | Control - Czech Republic | Computer Screen & Brief Physician Advice - Czech Republic
Serious Adverse Events (participants affected / at risk) | 0/1068 | 0/1028 | 0/297 | 0/292
Other Adverse Events (participants affected / at risk) | 0/1068 | 0/1028 | 0/297 | 0/292

LIMITATIONS AND CAVEATS:
Use of non-randomized, asynchronous study design may have confounded results; 2 NE groups not equivalent in baseline substance use (but controlled for in analysis); self-report and interview-collected data prone to recall and social desirability bias

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No